CLINICAL TRIAL: NCT02125656
Title: Use of High Intensity Interval Training as a Strategy to Minimize the Insulin Resistance Observed in Sleep Deprivation
Acronym: HIIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Hanna Karen Moreira Antunes, Doctor, Federal University of São Paulo
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 475074/2011-4
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Insulin Resistance; Sleep Deprivation
MeSH Terms: conditions — Insulin Resistance; Sleep Deprivation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regular Sleep (No Intervention): A single night of regular sleep
- Sleep Deprivation (No Intervention): A single night of sleep deprivation
- HIIT + Regular Sleep (Experimental): 2 weeks of HIIT and after a single night of regular sleep.
  Interventions: Other: High Intensity Interval Training
- HIIT + Sleep Deprivation (Experimental): 2 weeks of HIIT and after a single night of sleep deprivation
  Interventions: Other: High Intensity Interval Training

INTERVENTIONS:
Other: High Intensity Interval Training — 6 sessions in 2 weeks (Monday, Wednesday and Friday). Each training session will consist of repeated high-intensity efforts in a workload that matches the peak oxygen uptake for 60 seconds. These sprints are interspersed with active recovery for 75 seconds on low intensity (30W). The training sessions will have three minutes of heating in 30W. There will be 8 shots in the first and second session, 10 shots in the third and fourth session and 12 shots in the fifth and sixth session.
  Arms: HIIT + Regular Sleep; HIIT + Sleep Deprivation

SUMMARY:
Sleep is an essential biological process for life and great value to functions such as learning, memory processing , cell and brain repair. Recently, new evidence points to the relationship between lack of sleep and carbohydrate metabolism , establishing a framework for insulin resistance observed in studies with restriction and sleep deprivation on several nights and in a single night . To reverse this process , one of the most effective strategies is physical exercise and part listed in the literature as a non-pharmacological tool for prevention and health promotion , as well as in the treatment of some diseases . However , the pace of modern society causes people to practice less physical exercise , lack of time being the main reason . In this scenario, the High Intensity Interval Training ( HIIT ) emerges as a powerful strategy that induces major changes optimizing the time spent on such activity. Considering the benefits of this mode , the purpose of this study is to investigate the effects of high-intensity interval training in the context of insulin resistance observed during sleep deprivation. Will be recruited 20 male volunteers, aged between 18 and 35 years old, healthy, with normal sleep duration equivalent to 7-8 hours / night, not smoking and regular eating habits. They will be submitted to a protocol of 6 sessions of high-intensity interval training for two weeks, and since the end period, sleep normally, or be deprived of sleep for 24 hours. Biochemical (thyroid hormones, cortisol, glucagon, free fatty acid, cholesterol, glucose and insulin) will be undertaken as well as evaluation of body composition by plethysmography, basal metabolic rate by indirect calorimetry and insulin sensitivity through Oral Glucose Tolerance Test (OGTT) before and after the training period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Recreationally Active
* Eutrophic
* Sleep Duration about 7-8 hours

Exclusion Criteria:

* No Smoking
* Without Sleep disorders
* Nondiabetic

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Blood Glucose | Change from Baseline in Blood Glucose at 2 weeks of high intensity interval training
  Oral Glucose Tolerance Test (OGTT) is performed after at least 8 hours of fasting overnight, by oral administration of standard dose of 75g anhydrous glucose dissolved in water (dextrose). The plasma glucose levels are fasting measured (before administration of glucose state) and 30, 60, 90, 120, 180 and 240 minutes after administration. Volunteers will be advised to follow the same eating patterns before testing.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge FT de Souza, Msc, Principal Investigator — Federal University of São Paulo